CLINICAL TRIAL: NCT04550897
Title: A Phase 1/2 Study With BM7PE Immunotoxin in Colorectal Cancer Patients With Metastatic Disease Who Are Refractory to or With Intolerance to Last Line of Standard Chemotherapy.
Brief Title: A Phase I/II Study With BM7PE Immunotoxin in Colorectal Cancer Patients
Acronym: BM7PE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Geir Olav Hjortland, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BM7PE
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Intolerance last line standard chemotherapy

STUDY DESIGN:
Intervention Model Description: Phase 1 study in colorectal cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BM7PE treatment (Experimental): The BM7PE treatment will be administered as a 20-minute i.v. infusion. The treatment is repeated after 2 weeks (day 15). The patients will be treated as in-patients and will stay at the hospital until toxicity have decreased to grade 2 and or plasma AST and or ALT levels has started to decrease. For at least a minimum of 3 days.
  The dose administered to the patient will be 2.5, 5.0, 7.5, 10.0, 15.0 and 20.0 μg/kg body weight.
  Interventions: Drug: BM7PE

INTERVENTIONS:
Drug: BM7PE — BM7PE immunotoxin is supplied as a liquid solution and is diluted in 0.9% saline to a total volume of 250 ml.

SUMMARY:
This phase 1/2 study will evaluate the safety, tolerance and dose of BM7PE treating patients with colorectal cancer who have progressed to standard cell therapy or cannot tolerate such therapy. The study starts as a phase 1 study with the aim of assessing the final dose for this group of patients. Based on the results, the study will continue into a phase 2. The phase 2 study aim to examine overall survival ≥ 9.3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma of colon or rectum
* Ambulatory with an ECOG performance status 0-1
* At least 18 years of age
* Progressive disease on or last line of standard chemotherapy or intolerance to further chemotherapy
* Laboratory values as the following: ANC, Platelets, Hb, Creatinine, Bilirubin, ASAT, ALAT, Albumin levels, INR
* Signed informed consent and expected cooperation of the patients for the treatment, and follow-up must be obtained and documented according to ICH GCP, and national/local regulations

Exclusion Criteria:

* History of prior metastatic disease the last 3 years
* History of CNS or bone metastases
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia
* Chemotherapy/radiation therapy or major surgery within the last 4 weeks before start of treatment
* Alcohol or drug abuse
* Any reason why, in the opinion of the investigator, the patient should not participate
* Has a known history of Human Immunodeficiency Virus (HIV)
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* Is pregnant or breastfeeding, or expecting to conceive or father children within the project duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events related to BM7PE | 30 days after last dose of BM7PE
  To characterize the safety and toxicity of BM7PE by register adverse event in accordance with CTCAE 5.0

SECONDARY OUTCOMES:
Efficacy of the BM7PE: Overall survival | Through study completion, an average of 1 year
  The Overall survival will be measured by death registration
Efficacy of the BM7PE: progression free survival | From date of first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The progression free survival will be measured by MR (RECIST 1.1)
Radiological response to BM7PE | From date of first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Will be measured by CT (RECIST 1.1) response rate

CONTACTS AND LOCATIONS:
Overall Officials: Geir O Hjortland, MDPhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No